CLINICAL TRIAL: NCT05542342
Title: Phase II, Open-Label Study of Preliminary Efficacy of Sitravatinib in Combination With Tislelizumab in Patients With Metastatic Uveal Melanoma With Liver Metastases.
Brief Title: Sitravatinib and Tislelizumab in Patients With Metastatic Uveal Melanoma With Liver Metastases.
Acronym: SITISVEAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español Multidisciplinar de Melanoma (Other)
Collaborators: Mirati Therapeutics Inc. (Industry); BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM2101; 2021-002474-99 (EudraCT Number)
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): Patients will receive Sitravatinib 100 mg orally once daily in combination with tislelizumab 200 mg IV once every 3 weeks until progression of disease, unacceptable toxicity, death, or consent withdrawal, whichever occurs first. Treatment may be continued after progression according to physician criteria (with previous consultation with Coordinating investigator) until patients no longer receive clinical benefit.
  Interventions: Drug: Tislelizumab; Drug: Sitravatinib Malate

INTERVENTIONS:
Drug: Tislelizumab — 200 mg IV once every 3 weeks
Drug: Sitravatinib Malate — 100 mg orally once daily

SUMMARY:
SITISVEAL stablish the hypothesis that treatment with Tislelizumab + Sitravatinib will increase the Objective Response Rate in patients with Metastatic Uveal Melanoma (mUM) with liver metastases, compared with the current standard of care.

This is a non-randomized, single arm, multicenter, phase II study of Sitravatinib in combination with Tislelizumab in subjects with metastatic uveal melanoma and liver metastases. After informed consent is obtained, subjects will enter in the Screening phase to assess eligibility criteria and perform a mandatory tumor biopsy. Upon meeting criteria, eligible subjects will be entered into the Treatment phase. Patients will receive Sitravatinib 100 mg orally once daily in combination with tislelizumab 200 mg IV once every 3 weeks until progression of disease, unacceptable toxicity, death, or consent withdrawal, whichever occurs first. Treatment may be continued after progression according to physician criteria (with previous consultation with Coordinating investigator) until patients no longer receive clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed metastatic uveal melanoma with measurable disease not eligible for curative therapy.
2. Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. Patients must have at least 1 biopsiable liver metastasis.
3. Patients who are human leucocites antigen (HLA)-A02:01 positive can have received one prior therapy with Tebentafusp for metastatic disease.
4. Patients must be 18 years of age or older at time of study entry.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
6. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations not performed according to normal practice. Patients must consent for liver metastasis biopsies donation at day 0 and day +42 since treatment initiation.
7. Adequate normal organ and marrow function as defined below:

   a) Haemoglobin ≥9.0 g/dL b) Absolute neutrophil count (ANC) >1.5 x 109/L (> 1500 per mm3) c) Platelet count ≥ 100 x 109/L (>75,000 per mm3) d) Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with Coordinating Investigator e) Both aspartate aminotrnsferase (AST) and alanine aminotransferase (ALT) must be < 5 x ULN.

   f) Creatinine clearance ⩾40 ml/min calculated by Cockcroft-Gault or another validated method g) Urine protein:creatinine ratio (UPC) ≤1 or ≤2+ proteinuria on 2 consecutive dipsticks taken no less than 1 week apart h) Subjects with 2+ proteinuria on dipstick must also have UPC < 0.5 on 2 consecutive samples.
8. Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and for 6 months after the last dose of Tislelizumab and/or Sitravatinib, and have a negative urine or serum pregnancy test ≤ 7 days before first administration of Tislelizumab and Sitravatinib. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   a) Amenorrheic for ≥1 year in the absence of chemotherapy and/or hormonal treatments b) Luteinizing hormone (LH) and/or follicle stimulating hormone and/or estradiol levels in the post-menopausal range c) Radiation induced oophorectomy with last menses >1 year ago d) Chemotherapy induced menopause with >1 year interval since last menses e) Surgical sterilization (bilateral oophorectomy or hysterectomy) f) Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy) g) Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
9. For both male and female patients/partners: Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study and for ≥ 6 months after the last dose of Tislelizumab and/or Sitravatinib. A sterile male is defined as:

   1. One for whom azoospermia has been previously demonstrated in a semen sample examination as definitive evidence of infertility.
   2. Males with known "low sperm counts" (consistent with "sub-fertility") are not to be considered sterile for purposes of this study.
10. Patient is willing and able to comply with the protocol procedures for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
11. Must have a life expectancy of at least 12 weeks
12. Subjects must be able to swallow and retain oral medications and be without clinically significant gastrointestinal illnesses that would preclude absorption of Sitravatinib.
13. Adequately controlled blood pressure (BP):

Systolic BP ≤140 mmHg and diastolic BP ≤90 mmHg in the presence or absence of a stable regimen of antihypertensive therapy.

Exclusion Criteria:

1. Patients with concomitant malignancy other than non-melanoma skin cancer, or superficial bladder cancer controlled with local treatment.
2. Previous treatment with targeted therapies and/or anti-angiogenic agents such as VEGFR, MEK, BRAF, ERK inhibitors, with the exception of Tebentafusp.
3. Previous treatment with immune checkpoint inhibitors, either anti-PD1/PD-L1 (Including Tislelizumab), anti-CTLA-4, or other treatments.
4. Presence of brain or leptomeningeal involvement unless previously treated, off steroids at least 2 weeks, and considered stable. Patients with untreated central nervous system (CNS) metastases and/or carcinomatous meningitis identified either on the baseline brain imaging [RECIST]) obtained during the screening period or identified prior to signing the ICF. Patients whose brain metastases have been treated may participate provided they show radiographic stability (defined as 2 brain images, both of which are obtained after treatment to the brain metastases. These imaging scans should both be obtained at least four weeks apart and show no evidence of intracranial progression). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable either, without the use of steroids, or are stable on a steroid dose of ≤10mg/day of prednisone or its equivalent and anticonvulsants, for at least 14 days prior to the start of treatment. Brain metastases will not be recorded as RECIST Target Lesions at baseline.
5. Patients weighing <30kg will be excluded from enrollment.
6. Participation in another clinical study with an investigational product during the last 4 weeks.
7. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
8. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤28 days prior to the first dose of study drug. If sufficient wash-out time has not occurred due to the schedule or Pharmacokinetic properties of an agent, a longer wash-out period will be required, as agreed by Sponsor designated Coordinating Investigator and Principal Investigator.
9. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Coordinating Investigator.
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with Tislelizumab may be included only after consultation with the Coordinating Investigator.
   3. Known toxicity on prior checkpoint inhibitor treatment:

      I) Grade ≥ 3 immune-related adverse event (AE) related to checkpoint inhibitors.

      II) Grade 2 immune-related AE associated with checkpoint inhibitor unless the AE resolved or was well III) controlled by withholding the checkpoint inhibitor and/or treatment with steroids, with the exception of prior colitis, myocarditis, and pneumonitis, which are exclusionary.

      CNS or ocular AE of any grade related to checkpoint inhibitors. Note: Patients with a prior endocrine AE are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
10. Any concurrent chemotherapy, investigational medicinal product (IMP), biologic, or hormonal therapy for cancer treatment different to Sitravatinib and/or Tislelizumab. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
11. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
12. Major surgery within a minimum of 4 weeks prior to inclusion; patients must have recovered from any effects of any major surgery prior to inclusion. Note: Local surgery of isolated lesions for palliative intent and minor surgeries performed to obtain biological material for the study (i.e. liver biopsy) are acceptable.
13. History of allogeneic organ transplantation.
14. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    3. Any chronic skin condition that does not require systemic therapy
    4. Patients without active disease in the last 5 years may be included but only after consultation with the Coordinating Investigator
    5. Patients with celiac disease controlled by diet alone
15. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled/malignant hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, compromise Sitravatinib absorption, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
16. History of another primary malignancy except for:

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IMP and of low potential risk for recurrence
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    3. Adequately treated carcinoma in situ without evidence of disease

       17 -History of active primary immunodeficiency.

18- Active infection including tuberculosis (TB) (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibodies are eligible only if polymerase chain reaction is negative for HCV RNA.

19- Current or prior use of immunosuppressive medication within 14 days before the first dose of Tislelizumab. The following are exceptions to this criterion:

a) Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection) b) Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent c) Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)

20- Receipt of live attenuated vaccine within 30 days prior to the first dose of IMP. Note: Patients, if enrolled, should not receive live vaccines whilst receiving IMP and up to 30 days after the last dose of IMP.

21- Female patients who are pregnant (confirmed with positive pregnancy test) or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 6 months after the last dose of Tislelizumab and/or Sitravatinib therapy.

22- History of severe allergic reaction attributed to Sitravatinib or a similar VEGFR inhibitor or known hypersensitivity to any component of Sitravatinib dose composition

23- Known allergy or hypersensitivity to Tislelizumab or Sitravatinib or any of the excipients.

24- History of gastrointestinal perforation. Subjects with a history of abdominal fistula will be eligible if:

a) the fistula has been surgically repaired, b) there is no evidence of fistula for at least 6 months prior to inclusion, and c) the subject is deemed to be at low risk of recurrent fistula in the opinion of the Investigator.

25- History of intra-abdominal abscess within 3 months prior to inclusion

26- Clinically significant signs and/or symptoms of bowel obstruction within 3 months prior to inclusion

27- Resting ECG with clinically significant abnormal findings. i.e. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart).

28- Subjects with any one or more of the following:

a)History of myocardial infarction within 6 months prior to inclusion; patients with a history of myocardial infarction within 6 to 12 months prior to inclusion may be allowed following assessment b) Unstable angina within 6 months prior to inclusion c) Known significant cardiac disease (New York Heart Association [NYHA] classification of III or IV).

d) Concomitant medication known to cause prolonged QT which cannot be discontinued or changed to a different medication prior to enrollment

29- Left ventricular ejection fraction < lower limit of normal (LLN) per institutional guidelines, or <55%, if threshold for normal is not otherwise specified by institutional guidelines, for patients with the following risk factors:

a) Prior or planned treatment with anthracyclines (ie, PLD) b) Prior treatment with trastuzumab c) Prior central thoracic radiation therapy (RT), including exposure of heart to therapeutic doses of ionizing RT d) History of myocardial infarction within 6 to 12 months prior to inclusion e) Prior history of other significant impaired cardiac function.

30- History of stroke or transient ischemic attack within 6 months prior to inclusion.

31- History of significant hemorrhage within 4 weeks of first dose date.

32- Patients with:

1. With uncontrolled diabetes or > Grade 1 laboratory test abnormalities in potassium, sodium, or corrected calcium despite standard medical management or ≥ Grade 3 hypoalbuminemia ≤ 14 days before
2. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage (recurrence ≤ 14 days after intervention)
3. History of interstitial lung disease, non-infectious pneumonitis or uncontrolled lung diseases including pulmonary fibrosis, or acute lung diseases. Patients with significantly impaired pulmonary function, or who require supplemental oxygen at baseline must undergo an assessment of pulmonary function at screening

   33- Evidence of any other disease, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that puts the subject at high risk for treatment-related complication.

   34- Prior enrollment or treatment in a previous Tislelizumab and/or Sitravatinib clinical study regardless of treatment arm assignment.

   35- Any serious medical condition or psychiatric illness that would interfere in understanding of the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Objective Response rate (ORR) | Throughout the study period, approximately 1 year per patient
  ORR is defined as the proportion of patients with at least one visit response of complete response (CR) or partial response (PR) that is confirmed at least 4 weeks later according to Response evaluation criteria in solid tumors (RECIST) version 1.1 criteria.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Throughout the study period, approximately 1 year per patient
  For this protocol, PFS is defined as the time from the first dose of study treatment until objective tumor progression according to RECIST 1.1 criteria or death, whichever occurs first.
Overall survival (OS) | Throughout the study period, approximately 1 year per patient
  Overall Survival is defined as the time from the first dose of study treatment until death from any cause. Those patients that do not present a death event or are lost to follow up will be censored at the date of the last contact.
Frequency of Adverse Reactions | Throughout the study period, approximately 1 year per patient
  Percentage of patients who experienced an adverse reaction

CONTACTS AND LOCATIONS:
Overall Officials: Josep Maria Piulats, M.D. Ph.D., Study Chair — ICO L´Hospitalet
Locations (4):
- Spain (4):
  - Hospital Universitario Virgen de la Macarena, Seville, Andalusia
  - Institut Catala Oncologia (ICO) L´Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario la Paz, Madrid, Madrid
  - Hospital General Universitario de Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No